CLINICAL TRIAL: NCT01468077
Title: Multicenter, Randomized, Parallel Group Study to Compare the Incidence of Tocilizumab Related Infusion Reactions in Patients With Moderate to Severe Active RA, When Infusion is Given Over 31 Minutes Compared to 1 Hour
Brief Title: A Study in Patients With Moderate to Severe Active Rheumatoid Arthritis Comparing Different Infusion Durations of RoActemra/Actemra (Tocilizumab) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27901
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (2):
- Tocilizumab, Normal Administration (Experimental): Tocilizumab 8 mg/kg infusion of 60 minutes duration every 4 weeks for 6 infusions (up to 24 weeks)
  Interventions: Drug: Tocilizumab
- Tocilizumab, Fast Administration (Experimental): Tocilizumab 8 mg/kg infusion of 31 minutes duration every 4 weeks for 6 infusions (up to 24 weeks). The first infusion was 1 hour. If an infusion reaction occurred during any treatment, 1 hour infusions were used for all subsequent infusions
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 8 mg/kg infusion
  Other Names: RoActemra; Actemra

SUMMARY:
This multi-center, randomized, parallel-group, active-controlled, open-label study will evaluate the safety and efficacy of a shortened RoActemra/Actemra (tocilizumab) infusion time compared to the normal infusion time. Patients will be randomized to 8 mg/kg RoActemra/Actemra infusion of 31 minutes every 4 weeks or to RoActemra/Actemra 8 mg/kg infusion of 60 minutes every 4 weeks. The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 18 years of age, inclusive
* Diagnosis of rheumatoid arthritis of at least 6 months duration
* Moderate to severe active rheumatoid arthritis (DAS28 >/=3.2)
* Patients received at least 1 disease-modifying anti-rheumatic drug (DMARD) and/or 1 or more TNFalfa-inhibitors over a period of at least 8 weeks

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned surgery within 6 months following randomization
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* Functional class IV (ACR criteria)
* History of severe allergic reaction to human, humanized or murine monoclonal antibodies
* Known active current or history of recurrent infection (including tuberculosis)
* Primary or secondary immunodeficiency (history of or currently active)
* Body weight >150 kg
* Previous treatment with any cell-depleting therapies
* Previous treatment with tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Denmark (7):
  - Aalborg
  - Frederiksberg
  - Hellerup
  - Holbæk
  - Odense
  - Silkeborg
  - Svendborg
- Reykjavik, Iceland

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab, Normal Administration: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenously (IV) over 60 minutes once every 4 weeks for a total of 6 infusions during the 24-week treatment period.
- Tocilizumab, Fast Administration: Participants received tocilizumab 8 mg/kg IV once every 4 weeks for a total of 6 infusions during the 24-week treatment period. The first infusion (Baseline) was given over 60 minutes, and over 31 minutes the following 5 infusions.
Period: Overall Study
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Started | 22 | 25
Completed | 18 | 22
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population: All participants enrolled in the study who had been randomly assigned to one of the two study treatments.
Groups:
- Tocilizumab, Normal Administration: Participants received tocilizumab 8 mg/kg IV over 60 minutes once every 4 weeks for a total of 6 infusions during the 24-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.8) | 59.8 (13.1) | 58.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Infusion Reaction
Description: An infusion reaction was defined as any adverse event (AE) that occurred during the infusion or during the 24 hours following the infusion and deemed possibly or probably related to tocilizumab.
Time Frame: Baseline (Day 1), and Weeks 4, 8, 12, 16, and 20
Population: Safety Analysis Set (SAS) Population: All randomized participants who received at least one infusion of tocilizumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 22 | 25
Percentage of Participants | 13.6 | 12.0
Statistical Analysis 1: Comparison: Tocilizumab, Normal Administration vs Tocilizumab, Fast Administration; Test type: Superiority or Other; Risk Difference (RD) = 0.0164, 95% CI 2-sided [-0.2685 to 0.2988] — The CI (confidence interval) is calculated by Exact method based on binomial distribution

2. Secondary Outcome: Percentage of Participants Discontinuing Tocilizumab in Response to an AE or a Serious Adverse Event (SAE)
Description: All occurrences of participants who received at least 1 infusion of tocilizumab and then stopped tocilizumab infusions due to an AE or SAE were analyzed.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 20, and 24
Population: SAS Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 22 | 25
Percentage of Participants | 9.0 | 8.0

3. Secondary Outcome: Percentage of Participants Discontinuing Tocilizumab for Other Reasons
Description: Participants that stopped the administration of tocilizumab and discontinued the study prematurely due to reasons other than an AE or SAE were analyzed.
Time Frame: Baseline and Weeks, 4, 8, 12, 16, 20, and 24
Population: SAS Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 22 | 25
Percentage of Participants | 9 | 4

4. Secondary Outcome: Percentage of Participants With Increased Liver Enzyme Values of Greater Than (>)1.5 Times, or >3 Times, or >5 Times Over the Upper Limit of Normal (ULN) by Visit Among Participants Who Completed All Visits
Description: Increased liver enzyme values defined as Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) values of >1.5 times, or >3 times, or >5 times over the ULN. Almost none of the participants had increased measurements of AST, thus only values of ALT were presented. None of the participants presented with increased values of ALT above 3 or 5 ULN at any of the visits.
  ITT Completers is defined as a subset of the participants in the ITT population who completed all study visits.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers with liver enzyme datasets for each analyzed visit
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 17 | 21
Percentage of Participants
  ALT>1.5 ULN, Week 4 | 12 | 5
  ALT>1.5 ULN, Week 8 | 6 | 10
  ALT>1.5 ULN, Week 12 | 6 | 5
  ALT>1.5 ULN, Week 16 | 6 | 10
  ALT>1.5 ULN, Week 20 | 12 | 5
  ALT>1.5 ULN, Week 24 | 24 | 5

5. Secondary Outcome: Percentage of Participants With Increased Lipid Values by Visit Among Participants Who Completed All Visits
Description: Increased levels of high density lipoproteins (HDL) equal to or greater than (≥)1.5 millimoles per liter (mmol/L), and low density lipoproteins (LDL) ≥4.1 mmol/L, and total cholesterol ≥5.1 mmol/L, are defined according to the Adult Treatment Panel III (ATP-III) guidelines.
Time Frame: Screening and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  High HDL (≥1.5 mmol/L), Screening | 44 | 46
  High HDL (≥1.5 mmol/L), Week 4 | 44 | 55
  High HDL (≥1.5 mmol/L), Week 8 | 50 | 36
  High HDL (≥1.5 mmol/L), Week 12 | 39 | 50
  High HDL (≥1.5 mmol/L), Week 16 | 44 | 41
  High HDL (≥1.5 mmol/L), Week 20 | 39 | 36
  High HDL (≥1.5 mmol/L), Week 24 | 44 | 46
  High LDL (≥4.1 mmol/L), Screening | 0 | 14
  High LDL (≥4.1 mmol/L), Week 4 | 11 | 27
  High LDL (≥4.1 mmol/L), Week 8 | 6 | 32
  High LDL (≥4.1 mmol/L), Week 12 | 6 | 36
  High LDL (≥4.1 mmol/L), Week 16 | 6 | 23
  High LDL (≥4.1 mmol/L), Week 20 | 11 | 32
  High LDL (≥4.1 mmol/L), Week 24 | 6 | 18
  High total cholesterol (≥5.1 mmol/L), Screening | 33 | 59
  High total cholesterol (≥5.1 mmol/L), Week 4 | 56 | 73
  High total cholesterol (≥5.1 mmol/L), Week 8 | 61 | 73
  High total cholesterol (≥5.1 mmol/L), Week 12 | 56 | 68
  High total cholesterol (≥5.1 mmol/L), Week 16 | 61 | 64
  High total cholesterol (≥5.1 mmol/L), Week 20 | 61 | 59
  High total cholesterol (≥5.1 mmol/L), Week 24 | 56 | 64

6. Secondary Outcome: Percentage of Participants With a Reduction of at Least 1.2 Points in Disease Activity Score Based on 28-Joint Count (DAS28) by Visit Among Participants Who Completed All Visits
Description: Improvement in Rheumatoid Arthritis (RA) disease activity was measured by the DAS28 score, which is an index combining measurements of swollen and tender joints, acute phase response High sensitivity C-Reactive Protein (hsCRP), and global assessment of disease activity by the participant. A clinically meaningful improvement was defined as a reduction of at least 1.2 units in the DAS28 score during the study period. A low disease activity was defined as a DAS28 score less than (<)3.2, and remission was defined as a DAS28 score <2.6.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 67 | 55
  Week 8 | 89 | 73
  Week 12 | 89 | 82
  Week 16 | 94 | 77
  Week 20 | 94 | 82
  Week 24 | 89 | 86

7. Secondary Outcome: Percentage of Participants Achieving a DAS28 Score Below 3.2 (Low Disease Activity) by Visit Among Participants Who Completed All Visits
Description: Improvement in RA disease activity was measured by the DAS28 score, which is an index combining measurements of swollen and tender joints, acute phase response hsCRP, and global assessment of disease activity by the participant. A clinically meaningful improvement was defined as a reduction of at least 1.2 units in the DAS28 score during the study period. A low disease activity was defined as a DAS28 score <3.2, and remission was defined as a DAS28 score <2.6.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 44 | 27
  Week 8 | 67 | 55
  Week 12 | 78 | 82
  Week 16 | 94 | 68
  Week 20 | 89 | 73
  Week 24 | 83 | 77

8. Secondary Outcome: Percentage of Participants Achieving a DAS28 Score Below 2.6 (Remission) by Visit Among Participants Who Completed All Visits
Description: as for outcome 7
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 22 | 9
  Week 8 | 28 | 36
  Week 12 | 50 | 73
  Week 16 | 78 | 46
  Week 20 | 72 | 59
  Week 24 | 61 | 55

9. Secondary Outcome: DAS28 Score by Visit Among Participants Who Completed All Visits
Description: as for outcome 7
Time Frame: Baseline, Weeks, 4, 8, 12, 16, 20, and 24
Population: ITT Completers; n = the number of participants analyzed for the given parameter at the specific visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
scores on a scale
  Baseline (n=18,21) | 5.0 (1.1) | 5.0 (0.9)
  Week 4 (n=18,21) | 3.3 (0.8) | 3.6 (1.0)
  Week 8 (n=18,22) | 2.9 (0.8) | 3.1 (1.2)
  Week 12 (n=18,22) | 2.6 (0.9) | 2.4 (1.0)
  Week 16 (n=18,21) | 2.3 (0.4) | 2.6 (1.0)
  Week 20 (n=18,22) | 2.3 (0.6) | 2.6 (0.9)
  Week 24 (n=18,22) | 2.3 (0.6) | 2.5 (1.0)

10. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Percent (%) Improvement (ACR20 Response) by Visit Among Participants Who Completed All Visits
Description: ACR20 response is defined as an improvement of ≥20% in swollen joint count (SJC; 66 joints) and tender joint count (TJC; 68 joints) as well as ≥20% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; Health Assessment Questionnaire - Disability Index (HAQ-DI); and acute phase reactive factors (Erythrocyte Sedimentation Rate [ESR] or C-Reactive Protein [CRP]).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 50 | 41
  Week 8 | 67 | 59
  Week 12 | 72 | 68
  Week 16 | 83 | 77
  Week 20 | 83 | 73
  Week 24 | 89 | 91

11. Secondary Outcome: Percentage of Participants Achieving ACR 50% Improvement (ACR50 Response) by Visit Among Participants Who Completed All Visits
Description: ACR50 response is defined as an improvement of ≥50% in SJC (66 joints) and TJC (68 joints) as well as ≥50% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; HAQ-DI; and acute phase reactive factors (ESR or CRP).
Time Frame: Weeks, 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 28 | 18
  Week 8 | 28 | 36
  Week 12 | 50 | 50
  Week 16 | 44 | 46
  Week 20 | 67 | 55
  Week 24 | 72 | 73

12. Secondary Outcome: Percentage of Participants Achieving ACR 70% Improvement (ACR70 Response) by Visit, Among Participants Who Completed All Visits
Description: ACR70 response is defined as an improvement of ≥70% in SJC (66 joints) and TJC (68 joints) as well as ≥70% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; HAQ-DI; and acute phase reactive factors (ESR or CRP).
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 11 | 5
  Week 8 | 17 | 23
  Week 12 | 22 | 36
  Week 16 | 11 | 27
  Week 20 | 22 | 18
  Week 24 | 22 | 36

13. Secondary Outcome: Percentage of Participants Achieving ACR 90% Improvement (ACR90 Response) by Visit Among Participants Who Completed All Visits
Description: ACR90 response is defined as an improvement of ≥90% in SJC (66 joints) and TJC (68 joints) as well as ≥90% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; HAQ-DI; and acute phase reactive factors (ESR or CRP).
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 0 | 0
  Week 8 | 0 | 9
  Week 12 | 0 | 14
  Week 16 | 0 | 0
  Week 20 | 6 | 5
  Week 24 | 6 | 9

14. Secondary Outcome: High Sensitivity C-Reactive Protein (hsCRP) Levels by Visit Among Participants Who Completed All Visits
Description: hsCRP is a marker for inflammation and is measured in milligrams per liter (mg/L). High levels of this protein indicate inflammation in diseases such as RA.
Time Frame: Screening, Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Completers
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
mg/L
  Screening | 22.8 (19.8) | 25.9 (36.0)
  Baseline | 23.5 (22.7) | 27.0 (32.1)
  Week 4 | 4.7 (6.6) | 3.1 (3.4)
  Week 8 | 3.3 (3.3) | 4.5 (3.8)
  Week 12 | 3.2 (3.4) | 2.6 (3.3)
  Week 16 | 2.8 (3.1) | 3.1 (3.3)
  Week 20 | 2.9 (3.0) | 3.0 (3.2)
  Week 24 | 3.2 (3.5) | 3.4 (3.6)

15. Secondary Outcome: Modified Health Assessment Questionnaire (M-HAQ) Score by Visit Among Participants Who Completed All Visits
Description: M-HAQ is a self-reported, valid assessment of functional disability in RA. Assessment based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. Scores range 0 to 3; without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3.
Time Frame: Baseline, Weeks 4, 8, 12, 20, and 24
Population: ITT Completers
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
scores on a scale
  Baseline | 1.29 (0.71) | 1.50 (0.74)
  Week 4 | 0.97 (0.64) | 1.10 (0.64)
  Week 8 | 0.79 (0.67) | 0.95 (0.68)
  Week 12 | 0.80 (0.70) | 0.98 (0.62)
  Week 16 | 0.82 (0.69) | 0.94 (0.69)
  Week 20 | 0.75 (0.61) | 1.05 (0.77)
  Week 24 | 0.68 (0.63) | 1.07 (0.82)

16. Secondary Outcome: Percentage of Participants With Improvement of at Least 0.22 Units in M-HAQ Compared to Baseline Per Visit Among Participants Who Completed All Visits
Description: as for outcome 15
Time Frame: Weeks 4, 8. 12, 20, and 24
Population: ITT Completers
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Number analyzed (Participants) | 18 | 22
Percentage of Participants
  Week 4 | 44.4 | 45.5
  Week 8 | 72.2 | 59.1
  Week 12 | 72.2 | 54.5
  Week 16 | 77.8 | 63.6
  Week 20 | 66.7 | 59.1
  Week 24 | 72.2 | 50.0

ADVERSE EVENTS:
Time Frame: Screening through Week 24 (or early withdrawal). For early withdrawal two follow-up visits occurred; at 4 weeks and at 12 weeks after the last infusion. A telephone call was sufficient for the last visit if laboratory procedures were not needed.
Description: SAS Population
Arm/Group | Tocilizumab, Normal Administration | Tocilizumab, Fast Administration
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/25
Other Adverse Events (participants affected / at risk) | 20/22 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab, Normal Administration (N=22) | Tocilizumab, Fast Administration (N=25)
Infective tenosynovitis (Infections and infestations) | 1 | 0
Lymphoma cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab, Normal Administration (N=22) | Tocilizumab, Fast Administration (N=25)
Nasopharyngitis (Infections and infestations) | 3 | 5
Rhinitis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 2 | 3
Pain (General disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 4
Headache (Nervous system disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 3
Skin infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Contusion (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Eye allergy (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infective tenosynovitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.